CLINICAL TRIAL: NCT00688896
Title: A 4-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study Evaluating the Efficacy and Safety of JTT-705 (300 mg or 600 mg) Versus Placebo in Combination With Pravastatin 40 mg in Patients With Type II Hyperlipidemia
Brief Title: Efficacy and Safety Study of JTT-705 in Combination With Pravastatin 40 mg in Patients With Type II Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Shoji Hoshino, DVM, Vice President, Clinical Development, Akros Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT705-X-02-001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Type II Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — dalcetrapib; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): JTT-705 600 mg and pravastatin 40 mg
  Interventions: Drug: JTT-705 600 mg and pravastatin 40 mg
- 2 (Experimental): JTT-705 300 mg and pravastatin 40 mg
  Interventions: Drug: JTT-705 300 mg and pravastatin 40 mg
- 3 (Placebo Comparator): Placebo and pravastatin 40 mg
  Interventions: Drug: Placebo and pravastatin 40 mg

INTERVENTIONS:
Drug: JTT-705 600 mg and pravastatin 40 mg — * JTT-705 300 mg tablets, 600 mg dose, 2 tablets, oral, once daily, immediately following breakfast and/or assessment
  * Pravastatin 40 mg tablets, 40 mg dose, one tablet, oral, once daily, at bedtime
  Arms: 1
Drug: JTT-705 300 mg and pravastatin 40 mg — * JTT-705 300 mg tablets, 300 mg dose, 1 tablet, oral, once daily, immediately following breakfast and/or assessment
  * Placebo tablets, one tablet, oral, once daily, immediately following breakfast and/or assessments
  * Pravastatin 40 mg tablets, 40 mg dose, one tablet, oral, once daily, at bedtime
  Arms: 2
Drug: Placebo and pravastatin 40 mg — * Placebo tablets, 2 tablets, oral, once daily, immediately following breakfast and/or assessments
  * Pravastatin 40 mg tablets, 40 mg dose, one tablet, oral, once daily, at bedtime
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effect of two dose levels of JTT-705 when co-administered with pravastatin 40 mg on HDL-C and LDL-C and the inhibition rate of CETP activity and to document short term safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients having lipid values as indicated below:
* HDL-C less than 1.6 mmol/L (60 mg/dL)
* TG less than 4.5 mmol/L (400 mg/dL)
* LDL more than 4.0 mmol/L (160 mg/dL)
* Patients with CHD or CHD risk equivalent
* Male and females between 18 and 65 years of age (female patients must be post-menopausal, surgically sterile or using an acceptable form of contraception)

Exclusion Criteria:

* Body Mass Index of ≥ 35 kg/m2
* Females that are pregnant or breast-feeding, and females of child bearing potential who are not using an effective method of contraception
* Concomitant use of medications identified in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2002-06; Primary Completion 2003-04 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
% change from baseline in HDL-C; inhibition of CETP activity | 4-weeks

SECONDARY OUTCOMES:
% change from baseline in LDL-C and TC/HDL-C | 4-weeks
Plasma concentration of JTT-705 | 4-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam, Amsterdam, Netherlands